CLINICAL TRIAL: NCT04117321
Title: Mother-infant Microbiota Transmission and Its Link to the Health of the Baby
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Francis KL Chan, Professor, Chinese University of Hong Kong
Other Study IDs: MOMmy study
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Gut Microbiome; Mother to Child Transmission
Keywords: Mommy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, stool, saliva, hair, nail, nasopharyngeal swab, skin swab, buccal swab, placenta, cord blood, low Vaginal swab and breast milk samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pregnant women: Women who are being pregnant and plan to give birth in local hospital. Pregnant women who plan to stay in the same local area for at least 7 years post-delivery.
- New Born Baby: new born baby of an enrolled pregnant woman.
- Father of new born baby: Biological father of an enrolled new born baby.

SUMMARY:
The human intestinal tract harbors a diverse and complex microbial community, known as gut microbiota, which is critical in sustaining physiology, metabolism, nutrition and immune function. Dysbiosis of gut microbiota has been linked with obesity, hyperglycemia, hyperlipidemia, inflammatory bowel disease and other chronic inflammatory diseases. Gut microbiota is affected by host genetic markup, diet and life style; and therefore varied by human races and geographical locations.

The development of gut microbiota starts before birth. The infant's microbiome can impact on human health in later life. The microbiome of pregnant women are associated with early-life microbiota of their offspring as well as growth, neurodevelopment and the development of allergic and neurocognitive disorders.

Early childhood, when the microbiota is less mature and more malleable, is a golden age for microbiota manipulation to prevent disease. Studying microbiota at this golden age also allow us to dissect the development of a faulty microbiota and identify therapeutic targets to reverse it and cure diseases that are already developed.

ELIGIBILITY:
Pregnant women

Inclusion Criteria:

1. Being pregnant
2. Plan to give birth in local hospital
3. Competent to provide informed consent (no mental illness or dementia, etc. that will hinder their ability to undertake informed consent)
4. Plan to stay in the same local area for at least 7 years post-delivery Exclusion Criteria: No

New Born Baby Inclusion Criteria

1. Be a new born baby of an enrolled pregnant woman
2. One of the parents or legal guardian is competent to provide informed consent (no mental illness or dementia, etc. that will hinder their ability to undertake informed consent) Exclusion Criteria: No

Father of new born baby Inclusion Criteria

1. Biological father of an enrolled new born baby
2. Competent to provide informed consent (no mental illness or dementia, etc. that will hinder their ability to undertake informed consent) Exclusion Criteria: No

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This project will consist of a total 100,000 mother-baby pairs from all centers in 7 years. The study is exploratory in nature. In considering the number of events required for reliable quantification of different factors on a range of diseases, we decided to include 100,000 mother-baby pairs.
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2019-09-23 (Actual); Primary Completion 2026-10-02 (Estimated); Study Completion 2027-10-02 (Estimated)

PRIMARY OUTCOMES:
Develop a 100,000 pair of mother-baby longitudinal cohort | 8 year
  Set up a large scale database to collect data such as comprehensive clinical data, such as mother's and father's demographic and clinical information (e.g. age, weight, gender, family medical history, dietary, drug usage etc.)

SECONDARY OUTCOMES:
Dissect the important microbiome that maintain health | 8 year
  Study samples will be collected to characterize which microbiota will be transmitted from mother to baby by performing metagenomics of gut microbiome in stool and other samples
Seize the golden period of early life for prevention of human diseases | 8 year
  Study samples will be collected to characterize which microbiota induces disease by performing metagenomics of gut microbiome in stool and other samples and develop treatment with microbiota.

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong, China